CLINICAL TRIAL: NCT01319110
Title: Coenzyme Q10 in Post-Cardiac Arrest Cerebral Resuscitation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael N. Cocchi, MD, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010P000362
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Cardiac Arrest; Sudden Cardiac Arrest
Keywords: Cardiac Arrest; Post Cardiac Arrest; CoQ10; Ubiquinone; Post Arrest
MeSH Terms: conditions — Heart Arrest; Death, Sudden, Cardiac | interventions — coenzyme Q10; Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CoenzymeQ10 (Experimental): Patients will receive CoenzymeQ10 200mg three times per day for 7 days, until return to baseline neurologic status, or until death/discharge (whichever comes first). CoQ10 will be given through pre-existing NG or OG tube, and mixed with 20 ml of chocolate Ensure so as to blind investigators and staff.
  Interventions: Drug: Coenzyme Q10
- Placebo (Placebo Comparator): Patients will receive 20 ml chocolate Ensure (as a placebo) three times per day for 7 days, until return to baseline neurologic status, or until death/discharge (whichever comes first). Placebo will be given through pre-existing NG or OG tube.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Coenzyme Q10 — Patients will receive CoQ10 200mg three times per day for 7 days, until return to baseline neurologic status, or until death/discharge (whichever comes first). CoQ10 will be given through pre-existing NG or OG tube, and mixed with 20 ml of chocolate Ensure so as to blind investigators and staff.
  Other Names: Ubiquinone
  Arms: CoenzymeQ10
Dietary Supplement: Placebo — Patients will be given Chocolate Ensure via NG/ OG 3x daily as a placebo.
  Arms: Placebo

SUMMARY:
Specific Aim #1: To determine if levels of CoQ10 are low post-cardiac arrest (CA). We will perform a prospective trial with the primary endpoint of describing the prevalence of low serum CoQ10 levels.

Specific Aim #2: To determine if CoQ10 levels in post-CA patients can be increased with the administration of exogenous CoQ10.. We will perform a randomized control trial (RCT) of post-CA patients with the secondary endpoint of comparing CoQ10 levels among those randomized to CoQ10 supplementation vs placebo.

DETAILED DESCRIPTION:
Cardiac arrest (CA) occurs in nearly 350,000 patients in the U.S. each year with an estimated mortality of 60% in those surviving the initial arrest. Moreover, the overall prognosis for survivors is often limited by neurologic injury. Two randomized control trials (RCTs) have demonstrated that therapeutic hypothermia (TH) after CA improves survival and reduces neurologic morbidity. As a result of these studies, TH has become the standard of care in post-CA patients. The mechanism of action for TH is hypothesized to be a reduction in cerebral oxygen consumption that occurs following an ischemia-reperfusion injury. Another similar potential target following ischemia-reperfusion injury is mitochondrial function in the injured brain cells and attenuation of potentially damaging oxygen-free radicals. Specifically, optimizing mitochondrial function and reducing oxygen free radicals may enhance cellular function and mitigate cellular injury thereby leading to improved neurologic outcomes. Coenzyme Q10 (CoQ10) is an essential mitochondrial co-factor and free radical scavenger that has been found to have neuroprotective effects in various neurodegenerative disorders such as Parkinson's disease and Huntington's disease. Whether CoQ10 can provide neuroprotection in acute ischemia-reperfusion injury remains less clear, but has been recognized by the American Heart Association as a potentially promising neuroprotective agent. We hypothesize that the administration of exogenous CoQ10 will raise serum concentrations of CoQ10 and as such may mitigate the adverse effects of the post-CA ischemia-reperfusion injury on the brain by optimizing mitochondrial function and reducing oxygen-free radicals. We support this hypothesis by the following:

1. Ischemia-reperfusion injury disrupts normal mitochondrial function and increases O2 free radicals.
2. CoQ10 has been found to attenuate the effects of ischemia-reperfusion injury through optimizing mitochondrial function and mitigation of cellular apoptosis.
3. CoQ10 has neuroprotective effects in other neurodegenerative disorders.
4. Our group has unpublished preliminary data showing low CoQ10 levels in a majority of patients with septic shock, and that lower CoQ10 levels are significantly associated with multiple markers of the inflammatory cascade.
5. A pilot human trial in post-CA patients demonstrated a reduction in mortality and trend toward reduction in neurologic morbidity.

To test our hypothesis, we propose the following pilot study as proof of concept in preparation for a larger multicenter trial powered toward neurologic outcome and mortality. This pilot study will allow for a more informed power analysis for a larger trial, provide proof of concept for enrollment and administration of therapy, examine the time-frame for drug absorption into serum, and evaluate for tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age > 18 years)
2. Comatose after CA with subsequent return of spontaneous circulation

Exclusion Criteria:

1. Comatose status prior to CA
2. CoQ10 therapy within one month prior to CA
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Cocchi, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- See also: Beth Israel Deaconess Medical Center Cardiac Arrest Center — http://www.bidmc.org/cardiacarrestcenter

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CoenzymeQ10 | Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CoenzymeQ10 | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Low Serum CoQ10 Levels in Cardiac Arrest Patients
Description: The primary outcome will be describing the prevalence of low serum CoQ10 levels compared to standard laboratory control values.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CoenzymeQ10 | Placebo
Number analyzed (Participants) | 5 | 5
ug/mL | 0.706 (0.290137) | 0.66 (0.267955)

2. Secondary Outcome: Comparison of Serum CoQ10 Levels Randomized to Supplementation vs. Placebo
Description: The secondary outcome will be to compare serum CoQ10 levels among those post-arrest patients randomized to CoQ10 supplementation vs placebo.
Time Frame: 1 year
Population: This data was not collected when the study was performed
Arm/Group | CoenzymeQ10 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | CoenzymeQ10 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/5
Other Adverse Events (participants affected / at risk) | 1/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoenzymeQ10 (N=5) | Placebo (N=5)
Death (General disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoenzymeQ10 (N=5) | Placebo (N=5)
Gut suctioning (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes